CLINICAL TRIAL: NCT03249571
Title: Influence of 2-Weeks Flavonoid Supplementation and an Acute 45-Minute Walking Bout or 2.5-h Running Bout on Plasma Levels of Gut-Derived Phenolics
Brief Title: Flavonoids, Exercise, Gut-Derived Phenolics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: Reoxcyn Discoveries Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-0240
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-08

CONDITIONS: Exercise and Gut-derived Phenolics
Keywords: exercise; flavonoids; gut permeability; gut-derived phenolics
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized, parallel group design
Who Masked: Participant, Investigator
Masking Description: Flavonoid or placebo in capsules
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flavonoid (Experimental): Flavonoid supplement
  Interventions: Dietary Supplement: Flavonoid supplement
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Flavonoid supplement — 2-weeks ingestion of flavonoid supplement
  Arms: Flavonoid
Dietary Supplement: Placebo — 2-week ingestion of placebo supplement
  Arms: Placebo

SUMMARY:
PURPOSE:

1. PRIMARY: Using a randomized, parallel group design, this investigation will determine if the combination of 2-weeks polyphenol supplementation (using the Reoxcyn flavonoid supplement in capsule form) and one acute 45-minute brisk walking bout enhances the translocation of gut-derived phenolics into the circulation. A comparator group of runners (N=20) ingesting the flavonoid supplement for two weeks will be included (2.5 h run, 70% VO2max).
2. SECONDARY: Data from this study will determine if 2-weeks supplementation of the Reoxcyn flavonoid supplement is a sufficient time period to increase circulating levels of gut-derived phenolics, extending data collected from the previous 12-week community trial.

HYPOTHESIS: We hypothesize that an acute 45-minute brisk walking exercise bout (60% VO2max) following 2 weeks of increased polyphenol intake will be a sufficient exercise stimulus to increase gut permeability and the movement of gut-derived phenolics into circulation. If this hypothesis is confirmed, these data would have broad public health appeal, demonstrating that the combination of brisk walking and increased polyphenol intake augments circulating levels of health-restoring small phenolic molecules derived from bacterial breakdown in the colon.

DETAILED DESCRIPTION:
Research Design: Study participants (N=85) will be entered into the study and randomized to the flavonoid or placebo supplement groups for 2 weeks, with these two independent groups run in parallel (with N=80 anticipated to successfully complete all study phases). Supplements will be administered in a double-blinded manner in capsule form. Study participants will report to the research facility for baseline testing and orientation, and then pre-study and after 2-weeks supplementation, and then again 24 hour later. Four blood samples will be collected as shown in the Figure (pre- and post-supplementation, post-exercise/rest, and 24-hour post-exercise/rest). When reporting to the lab after 2-weeks supplementation, study participants will be randomized to either sit or walk briskly on treadmills for 45 minutes. A comparator group of 20 runners ingesting the flavonoid supplement and running 2.5 h in the lab will be included to allow a comparison between moderate and intense exertion (and to provide pilot data for a future study). Baseline Testing: One to two weeks before the start of the study, study participants (walkers and runner) will be given an orientation to the study and then provide voluntary consent. Instructions will be given for recording all food and beverage intake in 3-day food logs (Thursday, Friday, and Saturday prior to starting supplementation). Demographic and training histories will be acquired with questionnaires. Height, body weight, and percent body fat (seca Medical Body Composition Analyzer 514 bioelectrical impedance scale, Hanover, MD) will be measured. VO2max will be assessed using the Bruce's treadmill protocol, with oxygen consumption and ventilation continuously monitored using the Cosmed CPET metabolic system.

Pre-Supplementation Lab Visit: On the first day of the study, participants (walkers and runners) will return to the lab in a fasted state (9 or more hours with no food or beverage other than water). Blood samples will be taken from an antecubital vein with subjects in the seated position. Participants (walkers) will be given a 2-week supply of flavonoid or placebo capsules organized into supplement trays to facilitate compliance. Runners will be given a 2-week supply of flavonoid capsules. The 3-day food record will be reviewed and collected by the research team, and analyzed for nutrient and flavonoid content using the Food Processor v. 11.1 (ESHA Research, Salem, OR). Each food/beverage will be assessed for macro- and micro-nutrients, total flavonoids and subtotals for each of the six flavonoid subclasses, and two individual flavonoid values (quercetin, EGCG). During the 2-day period prior to visit #3 to the lab, and during the entire day that includes visit #3, participants will be asked to avoid food and beverages containing sucralose (Splenda) and mannitol. To avoid sucralose and mannitol, participants will be asked to check ingredient lists for diet sodas, yogurt and other dairy products, snack foods, chewing gum and candy, low-sugar products, toothpaste, and mouthwash.

Post-Supplementation Lab Visits:

After the 2-week supplementation period, participants (walkers and runners) will return to the lab in an overnight fasted state (on the same day of the week as the pre-supplementation lab visit).

Participants will turn in the supplement tray to verify compliance with ingesting the capsules. A blood sample will be collected. Participants (walkers) will be randomized to either sit for 45 minutes in the lab or to walk briskly for 45 minutes on a 5% graded treadmill at 60% VO2max (with metabolic monitoring during the first 5 minutes, and then at 15, 30, and 45 minutes) using the Cosmed CPET metabolic cart. Runners will run at 70% VO2max on an ungraded treadmill for 2.5 h, with metabolic measurements made every 30 minutes. Water will be given ad libitum for all participants, with no other beverage or food allowed. Just prior to the sitting or walking lab sessions, and the 2.5 h run, participants will consume a 150-ml solution containing 1 g sucrose, 1 g lactulose, 0.5 g L-rhamnose, 1 g erythritol, 1 g sucralose, 0.5 g mannitol.

Urine will be collected in plastic containers for 24 h in two separate fractions: 0-5 h and 5-24 h. No eating or drinking (except tap water) will be allowed during the first 5-h urine collection. Participants will return the next morning in an overnight fasted state, provide a blood sample, and turn in urine samples.

Urine collection guidelines to the subjects:

* You should collect every drop of urine during each collection period (5 hours from the start of the exercise bout, and then the second collection lasting to the next morning or 5 to 24 h from the start of exercise). It does not matter how much or little urine is passed each time, as long as every drop is collected.
* Collect every drop of urine during the day and night in the two collection bottles (0-5 hours, 5-24 hours, beginning with the start of the lab exercise test session). Store the bottles in the refrigerator. Be sure to collect any urine passed during bowel movements.
* Finish by collecting the first urine passed the next morning, adding it to the collection bottle. Bring both urine collection bottles with you to the lab (i.e., the morning after the exercise session when you will provide your final blood sample).

Flavonoid Supplement: Supplement and placebo capsules will be prepared by Reoxcyn Innovation Group LLC (Salt Lake City, UT). (SEE supplementation information in attached file). Ingredients will be the same as tested in the community trial: vitamin C (as ascorbyl palmitate) (Green Wave Ingredients, La Mirada, CA), wild bilberry fruit extract (25% total anthocyanins) (FutureCeuticals, Momence, IL), green tea leaf extract (50% EGCG) (Watson Industries, Inc., Pomona, CA), quercetin aglycone (Novel Ingredients, East Hanover, NJ), caffeine (Creative Compounds, Scott City, MO), and omega 3 fatty acids (Novotech Nutraceuticals, Ventura, CA). Capsule fill ingredients and excipients include Nu-Flow 70R (from rice hulls), tapioca from cassava root, natural bamboo silica, marshmallow root. Placebo capsules will contain only the fill ingredients and excipients (without the active ingredients). The daily serving for the walkers will be 2 flavonoid or 2 placebo capsules. Two flavonoid capsules provides 329 mg flavonoids (American adult average, depending on the study, is 240 mg per day). The daily serving for the runners will be 4 flavonoid capsules (658 mg flavonoids). Participants will be given a 2-week supply of the either the flavonoid or placebo capsules, with instructions on how to consume daily in split doses (1 with breakfast and 1 with lunch, or double that amount for the runners). Study participants will be allowed to add one extra capsule per day to increase consumption if one or two days of taking the supplement are missed. Study participants will ingest 2 capsules (4 for the runners) just after providing the blood sample during the walk/rest (or run) lab session.

SUPPLEMENT CAPSULES will be TESTED for flavonoid content pre- and post-study by Dr. Mary Ann Lila (NCSU, Plants for Human Health Institute, NCRC).

Targeted Metabolomics Analysis:

Gut-derived phenolic metabolites will be purified from plasma by SPE using an automated platform and in-house 96-well SPE protocol (60mg, 3mL; Phenomenex) for extraction of 100 μL tissue. All analytes have been previously optimized for extraction efficiencies of between 80-100% recoveries with CV≤10%. Extracts will be separated and quantified via liquid chromatography tandem-MS/MS involving previously published and validated methodologies. Briefly, HPLC-ESI-MS/MS analysis will be performed using a SCIEX UPLC coupled 6500 + MS/MS-QTRAP™ equipped with an electrospray ionization (ESI) Turbo-V source (blood and fecal metabolites), with samples injected onto a Kinetex PFP column and mobile phase gradient consisted of 0.1% formic acid (v/v) in water (A) and 0.1% formic acid (v/v) in acetonitrile (B), and a 24 min separation time. The targeted metabolite analysis protocol has been optimized and validated to detect greater than 200 analytes which are quantified relative to authentic commercial and synthetic standards in our library, with putative Phase II conjugates identified using fragmentation profiling involving 3-5 unique transitions. This involves scanning over 1000 transitions corresponding to sulfate, glucuronide, methyl and glycine conjugates. This SMRM methodology was previously optimized for the Rexocyn treatment and provides a significantly more sensitive method than traditional multiple reaction monitoring (MRM) scanning procedures, as it permits monitoring a greater number of transitions per unit of time, in addition to allowing unique compound-dependent parameters to be utilized for each analyte, resulting in enhanced sensitivity. Finally, metabolites will be confirmed on the basis of retention time (using authentic and synthesized standards where possible) and three or more precursor-to-product ion transitions. Seven-point matrix-matched calibration curves ranging from 0 to 10 μM will be used for the analysis of flavonoids or from 0 to 50 μM for the analysis of phenolic metabolites.

Intestinal Permeability, Urine Lactulose/Rhamnose:

Urine sugar concentrations will be determined by high-pressure liquid chromatography. Sucrose in 0-5-h urine, lactulose/rhamnose (L/R) ratio in 0-5-h urine, and sucralose/erythritol (S/E) ratio in 5-24-h urine will be used as indicators for gastroduodenal, small and large intestine permeability, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Females and males, 18 to 50 years of age
* Body mass index <35 kg/m2 (i.e., not moderately or severely obese)
* Body weight of 100 pounds and greater
* Willing to consume during the study less than 5 servings/day fruits and vegetables, less than 2 cups/day coffee, and no green tea.
* Willing to avoid use of non-steroidal anti-inflammatory drugs (NSAIDs), and all dietary and herbal supplements for the 2-week study (and starting one week prior to the study).
* Walkers: Regular history of walking (>100 min/week totaling all walking, both short or long duration episodes) and capable of walking 45 min briskly on a treadmill
* Runners: History of participating in 10 km to 42.2 km races and capable of running for 2.5 h on a treadmill.
* Non-smoker.
* Generally healthy and without chronic disease including cardiovascular disease (e.g., heart disease, stroke), cancer, type 1 and 2 diabetes, rheumatoid arthritis.
* Willing to maintain normal physical activity and diet habits, and make no formal attempts to lose weight during the 2-week study.

Exclusion Criteria:

* Use of aspirin or non-steroidal anti-inflammatory drugs (NSAIDs) [e.g. ibuprofen (Advil, Motrin, Nuprin), naproxen (Aleve, Naprosyn), and COX-2 inhibitors (Celebrex)] within one week prior to the study, and/or intent to use these drugs during the 2-week period of the study.
* Regular use of fish oil supplements, omega 3 supplements, or omega 3-based drugs (Lovaza, etc.) during the past one to two weeks and plans to use these supplements during the study.
* Pregnant or breastfeeding.
* Currently on a weight reducing plan or using weight-loss medications (e.g., selective serotonin reuptake inhibitors, steroids, Ritalin, appetite suppressors, Xenical, Diethylpropion), and plans to continue during the 2-week period of the study.
* Regular use of large dose nutrient, herbal, and dietary supplements during the past one to two weeks, and plans to use these during the 2-week period of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2017-08-29 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Plasma gut-derived phenolics | Pre- and post-2 weeks supplementation, post-exercise, 24-h post-exercise
  Biotransformed flavonoids by gut bacteria after ingestion

SECONDARY OUTCOMES:
Urine sugars | 24 h urine collection
  Gut permeability test, with measurement of ingested sugars in urine

CONTACTS AND LOCATIONS:
Overall Officials: David C. Nieman, DrPH, Principal Investigator — Appalachian State Univ
Locations (1):
- North Carolina Research Campus, Human Performance Lab, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No